CLINICAL TRIAL: NCT02319135
Title: A PHASE III, MULTICENTRE, RANDOMIZED, OPEN LABEL CLINICAL TRIAL OF AZACYTIDINE (VIDAZA®) VERSUS FLUDARABINE AND CYTARABINE (FLUGA SCHEME) IN ELDERLY PATIENTS WITH NEWLY DIAGNOSED ACUTE MYELOID LEUKEMIA.
Brief Title: Azacytidine (Vidaza®) Versus Fludarabine and Cytarabine (Fluga Scheme) in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia
Acronym: FLUGAZA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Dynamic Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLUGAZA
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine; Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fludarabine cytarabine (Active Comparator): Priming with daily administration of subcutaneous G-CSF (lenograstim or filgrastim 5 mcg /kg / day, days -1, 1 and 2) (not given if hyperleukocytosis> 25 x 109/l), followed by:
  * Oral fludarabine (40 mg/m2/day, days 1 to 5) and subcutaneous cytarabine (75mg/m2/day, days 1 to 5) (FLUGA scheme) (fludarabine and cytarabine only days 1 to 4 if age ≥75 years), OR
  * Fludarabine (25 mg/m2/day) and cytarabine (75 mg/m2/day infusion of 6 hours) on their intravenous formulations if the patient is hospitalized (patients with hyperleukocytosis or other unfavourable conditions).
  Treatment cycles every 28 days
  Interventions: Drug: Fludarabine; Drug: Cytarabine; Drug: Lenograstim; Drug: Filgastrim
- Azacitidine (Experimental): Subcutaneous Azacitidine 75 mg/m2/day, days 1 to 7. Treatment cycles every 28 days.
  Interventions: Drug: Azacitadine

INTERVENTIONS:
Drug: Azacitadine
  Arms: Azacitidine
Drug: Fludarabine
  Arms: fludarabine cytarabine
Drug: Cytarabine
  Arms: fludarabine cytarabine
Drug: Lenograstim
  Arms: fludarabine cytarabine
Drug: Filgastrim
  Arms: fludarabine cytarabine

SUMMARY:
The hypothesis is that the replacement of the standard fludarabine and cytarabine based therapy by azacytidine could result in an improvement of RFS and OS rates in the experimental arm. To fulfill the medical needs in such frail and elderly population, improvements in terms of atileukemic efficacy in the azacytidine experimental arm should be attained without increasing the therapy-related toxicity or decreasing the patients QoL.

DETAILED DESCRIPTION:
This is a multicenter, randomized 1:1, open, and at national level, Phase III clinical trial.

This study will be conducted in 3 phases of different duration:

1. Selection phase (up to 14 days from the signature of informed consent): informed consent and review of the inclusion and exclusion criteria performing the relevant assessments.
2. Treatment Phase (from the start of treatment until the end of cycle 9): Induction phase (3 cycles) and consolidation phase (cycles 4-9). Study visits during treatment will be weekly during the induction phase (first 3 cycles) and every 2 weeks until the end of the consolidation phase.
3. Follow-up phase: monthly monitoring will be performed on all patients until they have completed a minimum of 2 years from the start of treatment, whether or not they continue receiving azacitidine cycles or Mini-Fluga according to the protocol. Following these 24 months, follow-up will be carried out at least quarterly. Patients suffering disease progression or relapse of the disease, or being early withdrawn due to any of the reasons specified in the protocol will be followed-up for survival until the end of the study or until the death of all patients, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. - Having voluntarily given informed consent before performing any test that is not part of

   routine care of patients.
2. - Age greater than or equal to 65.
3. - Morphological diagnosis of non-promyelocytic AML according to the WHO criteria.
4. - Newly diagnosed AML.
5. - ECOG performance status <4.
6. - Ability and willingness to comply with the schedule of study visits.

Exclusion Criteria:

1. - Genetic diagnosis of acute promyelocytic leukemia.
2. - Patients with AML secondary to myelodysplastic syndrome (MDS) or chronic myeloproloferative syndrome who have been previously treated with antileukemic agents

   (hypomethylating or standard chemotherapy). Treatment with hydroxyurea prior to randomization is allowed.
3. - Serum creatinine ≥ 250 mmol / l (≥ 2.5 mg/dL) (unless attributed to AML).
4. - Bilirubin, alkaline phosphatase or ALT > 5 times the value of the upper limit of normal (unless attributed to AML) .
5. - Presence of an active and/or non controlled pathology different to AML which is severe and life-threatening, that in the investigator's opinion, prevents the subject participation in the study.
6. - Other active concomitant malignancy or whose remission is less than one year from the screening day (except carcinoma in situ).
7. - Presence of any psychiatric illness or medical condition that, in the investigator's opinion, prevents the subject participation in the study.
8. - Life expectancy less than X months.
9. - Inability of the patient or his legal representative to understand and voluntarily sign the informed consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 289 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Efficacy (overall survival (OS) attained without increasing the therapy-related toxicity or decreasing the patients QoL. | 4 years
  To evaluate the overall survival (OS) in one year treatment with 2 first-line regimens in newly diagnosed elderly patients: 3 cycles of induction chemotherapy based on fludarabine and cytarabine (FLUGA scheme) followed by maintenance with reduced doses(Mini-FLUGA) (standard treatment arm) versus subcutaneous azacitidine cycles (experimental treatment arm).

SECONDARY OUTCOMES:
Efficacy (Event free survival (EFS) | 4 years
  Event free survival (EFS)
Efficacy (Duration of remission.) | 4 years
  Duration of remission.
Efficacy (Overall survival) Efficcacy | 3 years
  Overall survival at 2nd and 3rd year.
Safety (Compare hematologic and non-hematologic toxicity) | 3 years
  Compare hematologic and non-hematologic toxicity in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, Dr, Principal Investigator — PETHEMA Foundation
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Spain

REFERENCES:
- [Derived] Ayala R, Rapado I, Onecha E, Martinez-Cuadron D, Carreno-Tarragona G, Bergua JM, Vives S, Algarra JL, Tormo M, Martinez P, Serrano J, Herrera P, Ramos F, Salamero O, Lavilla E, Gil C, Lopez Lorenzo JL, Vidriales MB, Labrador J, Falantes JF, Sayas MJ, Paiva B, Barragan E, Prosper F, Sanz MA, Martinez-Lopez J, Montesinos P, On Behalf Of The Programa Para El Estudio de la Terapeutica En Hemopatias Malignas Pethema Cooperative Study Group. The Mutational Landscape of Acute Myeloid Leukaemia Predicts Responses and Outcomes in Elderly Patients from the PETHEMA-FLUGAZA Phase 3 Clinical Trial. Cancers (Basel). 2021 May 18;13(10):2458. doi: 10.3390/cancers13102458. PMID 34070172
- See also: CRO — http://www.dynasolutions.com